CLINICAL TRIAL: NCT01152086
Title: The Effects of Regular Mountain Hiking on Hopelessness in Chronically Suicidal Patients
Acronym: MOHS2010
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Prof. Josef Niebauer M.D., Ph.D., Prim. Prof. MD, PhD, MBA, Paracelsus Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hiking2010
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Suicide; Hopelessness
Keywords: Physical activity; mountain hiking; exercise; training program; hopelessness; chronic suicidality; depression; suicide attempt; suicide
MeSH Terms: conditions — Suicide; Motor Activity; Depression; Suicide, Attempted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hiking first (Active Comparator): This group first starts with mountain hiking over 9 weeks followed by a 9 weeks control period.
  Interventions: Other: Mountain hiking in the Austrian and Bavarian Alps
- Control first (Active Comparator): This group first starts with the control period (9 weeks) followed by the 9 weeks mountain hiking intervention.
  Interventions: Other: Mountain hiking in the Austrian and Bavarian Alps

INTERVENTIONS:
Other: Mountain hiking in the Austrian and Bavarian Alps — Regularly supervised physical exercise training program.
  Duration over all: 9 weeks; Frequency: 2 times per week; Duration one training-unit: 3 hours;
  Program:
  * Endurance training (performed within 70-85% of the maximum heart rate)
  * Short exercises before hiking (Mobilisation, Body and nature perception, ca. 5 min)
  * Stretching after hiking (ca. 5 min)
  * Short break at half-time (ca. 15 min)

SUMMARY:
Suicide is a major public health issue with estimated 1 million deaths worldwide within the last year. Physical activity and nature recreation might be protective factors against suicidal behaviour, suicidal ideation and contributing factors like depression and hopelessness.

In this randomized controlled cross-over intervention study the investigators aim to investigate the physical and psychological effects of a 9 weeks hiking program in chronically suicidal patients. The investigators aim to enroll 24 patients suffering from chronic suicidality, defined as at least one attempted suicide and a hopelessness greater than 26 in Beck's Hopelessness Scale summary score. At baseline patients will undergo pre-tests including questionnaires to assess suicide ideation, hopelessness, depression, anxiety, quality of life and health-related physical activity, physiological investigations to assess exercise capacity and blood investigations. Randomly assigned 12 patients start with the 9 weeks supervised mountain hiking program followed by a 9-week-period without supervised exercise program. The other 12 patients start with 9 weeks without supervised exercise program followed by a 9-week-period of supervised mountain hiking program. The mountain hiking program includes 2 training sessions per week with a duration of 3 hours per session. The hiking intervention will be performed within 70-85% of heart rate reserve and gymnastics for body and nature perception, mobilisation and stretching will enrich the training program. Further investigations including questionnaire-assessments, assessment of exercise capacity and blood investigations will be scheduled 9 and 18 weeks after the study start. In addition a daily assessment of several suicide risk-factors based on a web-based questionnaire will be done over the full study period. Within this mountain hiking program the investigators hope to reduce hopelessness in chronically suicidal patients.

ELIGIBILITY:
Inclusion Criteria:

Chronically suicidal defined as:

* at least one attempted suicide
* BHS summary scale > 26

Exclusion Criteria:

* Coronary heart disease defined by angina pectoris or relevant ST-changes during exercise or myocardial infarction in the last 6 months
* not oriented in time and space
* demented
* acute psychotic
* cognitively impaired
* insufficient german language skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Hopelessness | 18 weeks (3 time points)
  Summary score BHS (Beck Hopelessness Scale; 20 items)

SECONDARY OUTCOMES:
Exercise capacity | 18 weeks (3 time points)
  (Watts/kg)
Depression | 18 weeks (3 time points)
  BDI-2 summary score (Beck depression inventory 2, 21 items)
Anxiety | 18 weeks (3 time points)
  Summary score BAI (Beck anxiety inventory, 21 items)
Suicide ideation | 18 weeks (3 time points)
  Summary score BSI (Beck suicide ideation inventory, 21 items)
Quality of life | 18 weeks (3 time points)
  PLC (Profil der Lebensqualität Chronisch Kranker, 6 subscales: Leistungsvermögen, Genuß- und Entspannungsfähigkeit, Positive Stimmung, Negative Stimmung, Kontaktvermögen, Zugehörigkeitsgefühl)
Blood parameters of inflammation | 18 weeks (3 time points)
  Interleukin 1 beta, Interleukin 2, Interleukin 6, Interferon gamma, Interleukin 10, Interleukin 17;
suicide risk factors | 18 weeks (daily)
  Several items:
  * Grundwert aus dem Test zur existentiellen Motivation (Eckhard, 2000, 2 items)
  * Burdensomeness and Connectedness (Interpersonal needs questionnaire, Joiner 2005, 3 items)
  * Chronic Suicidality (Paris, 2007, 2 items)
  * Suicidal Status Form (SSF, Jobes, 2006, 9 items)
  * Emotionalität und Problembelastung (SNS-subscala, Schiepek, 9 items)
  * Alcohol consumption (1 item)
  * Sleep quality (1 item)
  * Social support (F-SozU-S54, 4 items)
  * Physical activity (IPAQ-short, 2 items)
  * Environmental perception (3 items)
  * Religiousness and spirituality (2 items)
health-related physical activity | 18 weeks (3 time points)
  IPAQ short version (International physical activity questionnaire, 2002)

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Fartacek, MD, MBA, Study Chair — Paracelsus Medical University

REFERENCES:
- [Background] Babiss LA, Gangwisch JE. Sports participation as a protective factor against depression and suicidal ideation in adolescents as mediated by self-esteem and social support. J Dev Behav Pediatr. 2009 Oct;30(5):376-84. doi: 10.1097/DBP.0b013e3181b33659. PMID 19692930
- [Background] Brown DR, Galuska DA, Zhang J, Eaton DK, Fulton JE, Lowry R, Maynard LM. Psychobiology and behavioral strategies. Physical activity, sport participation, and suicidal behavior: U.S. high school students. Med Sci Sports Exerc. 2007 Dec;39(12):2248-57. doi: 10.1249/mss.0b013e31815793a3. PMID 18046198
- [Background] Simon TR, Powell KE, Swann AC. Involvement in physical activity and risk for nearly lethal suicide attempts. Am J Prev Med. 2004 Nov;27(4):310-5. doi: 10.1016/j.amepre.2004.07.003. PMID 15488361
- [Background] Taliaferro LA, Rienzo BA, Pigg RM Jr, Miller MD, Dodd VJ. Associations between physical activity and reduced rates of hopelessness, depression, and suicidal behavior among college students. J Am Coll Health. 2009 Jan-Feb;57(4):427-36. doi: 10.3200/JACH.57.4.427-436. PMID 19114382
- [Background] Tao FB, Xu ML, Kim SD, Sun Y, Su PY, Huang K. Physical activity might not be the protective factor for health risk behaviours and psychopathological symptoms in adolescents. J Paediatr Child Health. 2007 Nov;43(11):762-7. doi: 10.1111/j.1440-1754.2007.01217.x. PMID 17924938